CLINICAL TRIAL: NCT06438107
Title: Deep Phenotyping of the Renal Allograft to Prognosticate Clinical Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Aravind Cherukuri, Assistant Professor of Medicine and Surgery, University of Pittsburgh
Other Study IDs: STUDY21090074
Record Dates: First submitted 2024-02-19; First posted 2024-05-31 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Renal Transplant Rejection
Keywords: Organ rejection; Acute rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Renal biopsy core tissue specimens, blood plasma and PBMC samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal transplantation recipients: Living donor and deceased donor renal transplant recipients. There is no intervention to be administered.

SUMMARY:
The goal of this observational study is to determine phenotypic, transcriptional, and epigenetic underpinnings of renal allograft rejection in renal transplant rejection. The main questions it aims to answer are:

* To determine the phenotype, frequency, location, and the inter-cellular interactions between the cells that constitute intra-graft inflammatory infiltrate in acute ejection.
* To determine the phenotype, frequency, location, and the inter-cellular interactions between the cells that constitute intra-graft inflammatory infiltrate in recurrent/recalcitrant rejection vs. rejection that resolves with therapy.
* To generate a scRNA sequencing (scRNAseq) map of the intra-graft immune cells and the renal parenchymal cells and compare the transcriptional and epigenetic changes within these cells in recurrent/recalcitrant rejection vs. rejection that resolves with therapy.
* To determine phenotypic changes associated with chronic rejection.

Participants will be asked to provide the following research specimens:

* Renal biopsy specimens at the following timepoints: day of transplantation (pre-implantation and post-perfusion); routine protocol biopsies at 3 months and 12 months; and clinically indicated for-cause biopsies at any timepoint from time-0 to 1-yr post-transplantation. The 1st research core will be used for routine histopathological examination and left over tissue from this core will be used for deep phenotyping using multiparameter immunophenotyping, and digital spatial profiling. The second research core will be used for extraction of cells and nuclei for scRNAseq and snATACseq.
* Blood samples will be processed to obtain plasma (for cytokine, chemokine and DSA measurements) and PBMC (for deep phenotyping and molecular analyses). For each collection timepoint, up to 75 mL (about 5 tablespoons) will be collected.
* Prospective clinical data and outcomes will be collected from participant medical records.
* Follow-Up Period: For-cause biopsies from 1-yr to 5-yr post-transplantation (by the transplant nephrologist): no additional cores will be obtained for research from these biopsies. The left-over tissue from the clinically indicated biopsy cores will be analyzed by deep phenotyping and digital spatial profiling. Blood samples will be processed to obtain plasma (for cytokine, chemokine and DSA measurements) and PBMC (for deep phenotyping and molecular analyses).

DETAILED DESCRIPTION:
This study is exploratory in nature and aims to elucidate the phenotypic, transcriptional, and epigenetic underpinnings of renal transplant rejection. The study is designed to provide improved understanding of the regulation of intra-graft alloimmune response in the renal transplant recipients.

In this single center, prospective, longitudinal, observational cohort study, sequential assessment of renal biopsies will be performed at baseline (pre-implantation), 3 months and at one-year post-transplantation in addition to any for-cause biopsies within the first five years post-transplantation. Blood samples will be also collected at the time of renal biopsies for comparison analyses.

HYPOTHESIS It is proposed that unique phenotypic, transcriptional, and epigenetic changes within the parenchymal and the infiltrating nonparenchymal inflammatory cells dictate the evolution of renal allograft inflammation and rejection.

The following research specimens will be obtained from each study participant:

1. The day of transplantation (by the UPMC operating surgeon): Pre-implantation core renal biopsy and post-perfusion core renal biopsy: Two research cores for each biopsy will be taken from the transplanted kidney. The pre-implantation biopsy specimens are obtained on the back table, and the post-perfusion cores are taken prior to closure of the surgical incision. The 1st research core will be used for routine histopathological examination and left over tissue from this core will be used for deep phenotyping using multiparameter immunophenotyping, and digital spatial profiling. The second research core will be used for extraction of cells and nuclei for scRNAseq and snATACseq. Blood samples will be processed to obtain plasma (for cytokine, chemokine and DSA measurements) and PBMC (for deep phenotyping and molecular analyses). For each collection timepoint, up to 75 mL (about 5 tablespoons) will be collected.
2. Protocol biopsies at 3 months and 12 months (by the transplant nephrologist): Renal transplant recipients at UPMC routinely undergo clinical post-transplant biopsies at 3 months and at 12 months. An additional research core will be collected along with the clinically indicated biopsy cores at both these time points (3 total passes of the biopsy needle for each collection). Left over tissue from the clinically indicated core will be used for deep phenotyping using multiparameter immunophenotyping, and digital spatial profiling. The research core will be used for extraction of cells and nuclei for scRNAseq and snATACseq. Blood samples will be processed to obtain plasma (for cytokine, chemokine and DSA measurements) and PBMC (for deep phenotyping and molecular analyses).
3. For-cause biopsies from time-0 to 1-yr post-transplantation (by the transplant nephrologist): Along with the protocol biopsies, UPMC renal transplant patients also undergo biopsies for clinical indication (for-cause biopsies). Again, an additional research core will be collected along with the clinically indicated biopsy cores whenever a patient undergoes any for-cause biopsy between time-0 and 1-year post-transplantation (3 total passes of the biopsy needle for each collection). Left over tissue from the clinically indicated core will be used for deep phenotyping using multiparameter immunophenotyping, and digital spatial profiling. The research core will be used for extraction of cells and nuclei for scRNAseq and snATACseq. Blood samples will be processed to obtain plasma (for cytokine, chemokine and DSA measurements) and PBMC (for deep phenotyping and molecular analyses).

The investigators will review procedures associated with the consent with participants again at the time of each of these biopsies to confirm their continued interest in participation. As these procedures are a part of the standard of care biopsies that the patients undergo, no additional hospital visits are expected. The research specimens will be delivered to and processed by laboratory research members.

Prospective clinical data and outcomes will be collected from participant medical records.

The following clinical data will be collected from each research participant:

1. Demographic characteristics (e.g., age, gender, ethnicity, cause of renal disease)
2. Pre-transplant clinical variables (e.g., h/o prior transplant, HLA mismatches, panel reactive antibodies, prior use of immunosuppression, cold ischemia time, warm ischemia time)
3. De-identified donor data (e.g., donor age, gender, ethnicity, donor type, KDPI) as available at time of transplant
4. Immunosuppression details (e.g., induction and maintenance agents, trough CNI levels through the 1st post-transplant year)
5. Clinical outcomes (e.g., DGF; detection of DSA; biopsy clinical reports; Serum Creatinine and eGFR at 1, 3, 6, and 12 months, and then at 2, 3, 4, and 5 years; graft and patient survival at 5 years)

Follow-Up Period For-cause biopsies from 1-yr to 5-yr post-transplantation (by the transplant nephrologist): These are the standard-of-care indication biopsies that are performed beyond the 1st post-transplant year, up to 5 years post-transplantation. While no additional cores will be obtained for research from these biopsies (about 2 passes of the biopsy needle per standard practices), we will analyze the left-over tissue from the clinically indicated biopsy cores by deep phenotyping (Marcus Clark Lab, University of Chicago; MTA in place) and digital spatial profiling (Randhawa Lab, University of Pittsburgh). Blood samples will be processed to obtain plasma (for cytokine, chemokine and DSA measurements) and PBMC (for deep phenotyping and molecular analyses).

STUDY AIMS Aim 1. To determine phenotypic, transcriptional, and epigenetic underpinnings of renal allograft rejection.

1. A) To determine the phenotype, frequency, location, and the inter-cellular interactions between the cells that constitute intra-graft inflammatory infiltrate in acute ejection. (1B) To generate a scRNA sequencing (scRNAseq) map of the intra-graft immune cells and the renal parenchymal cells and determine the transcriptional and epigenetic changes within these cells at baseline, prior to the diagnosis, and at the diagnosis of acute rejection. Analysis of these changes longitudinally through the 1st post-transplant year will allow us to delineate the natural history of renal allograft rejection.

   Aim 2. To determine phenotypic, transcriptional, and epigenetic differences that underlie persistence vs. resolution of acute rejection after renal transplantation.
2. A) To determine the phenotype, frequency, location, and the inter-cellular interactions between the cells that constitute intra-graft inflammatory infiltrate in recurrent/recalcitrant rejection vs. rejection that resolves with therapy. (2B) To generate a scRNA sequencing (scRNAseq) map of the intra-graft immune cells and the renal parenchymal cells and compare the transcriptional and epigenetic changes within these cells in recurrent/recalcitrant rejection vs. rejection that resolves with therapy.

Aim 3. To determine phenotypic changes associated with chronic rejection. In a subset of patient in whom for-cause transplant biopsies are available past the 1st year and up to 5 years after transplantation, we will perform multi-parameter immunophenotyping and spatial transcriptional analysis to explore cellular infiltrate and transcriptional changes associated with chronic rejection.

Exploratory Endpoints:

1. To correlate the frequency and phenotype of the intra-graft inflammatory infiltrate with histological diagnosis within the 1st post-transplant year (acute rejection vs. borderline rejection vs. no acute rejection).
2. To determine the transcriptional and epigenetic changes within intra-graft immune cells and graft parenchymal cells at baseline, prior to and at the diagnosis of acute rejection or borderline rejection in comparison to no rejection.
3. To determine phenotypic, transcriptional, and epigenetic differences that underlie persistence vs. resolution of acute rejection in the 1st post-transplant year.
4. To determine the phenotypic and transcriptional changes associated with chronic rejection.
5. To correlate histological phenotypes with peripheral blood phenotypes.

ELIGIBILITY:
Inclusion Criteria:

1. All adult living or deceased donor renal transplant recipients (age ≥ 18 years), irrespective of gender, race, or ethnic background.
2. Able to understand and provide inform consent.

Exclusion Criteria:

1. Medical contraindications to undergo renal biopsy (use of long-term anticoagulation, low platelet count of <100,000/uL)
2. Cause of ESRD likely to recur in transplant: Hemolytic uremic syndrome (HUS)
3. Not maintained on standard of care immunosuppression therapy (Thymoglobulin induction followed by tacrolimus and mycophenolate maintenance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult living donor or deceased donor renal transplant recipients
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Biopsy Proven Acute Rejection at one year | 1 year
  Percentage biopsy proven acute rejection either on a surveillance biopsy or a for-cause biopsy in the First Post-Transplant Year
Degree of Correlation of Acute Rejection Transcriptional Changes Within the Infiltrating Inflammatory Cells at one year | 1 year
  Degree of Correlation of Transcriptional Changes Within the Infiltrating Inflammatory Cells Assessed by scRNA Sequencing in the First Post-Transplant Year
Percentage of Correlation of Transcriptional Changes Within the Renal Parenchymal Cells at one year | 1 year
  Percentage Correlation of Acute Rejection Transcriptional Changes Within the Renal Parenchymal Cells Assessed by scRNA Sequencing in the First Post-Transplant Year

SECONDARY OUTCOMES:
Percentage of Histological Persistence of Rejection at one year | 1 year
  Percentage Histological Persistence of Rejection in the First Post-Transplant Year
Degree of Correlation of Histological Transcriptional Changes Within the Infiltrating Inflammatory Cells at one year | 1 Year
  Degree of Correlation of Histological Transcriptional Changes Within the Infiltrating Inflammatory Cells in the First Post-Transplant Year
Degree of Correlation of Histological Transcriptional Changes Within the Renal Parenchymal Cells at one year | 1 Year
  Degree of Correlation of Histological Transcriptional Changes Within the Renal Parenchymal Cells in the First Post-Transplant Year
Percentage of Participants with Biopsy Proven Acute Rejection at Year 3 | 3 Years
  Percentage biopsy proven acute rejection either on a surveillance biopsy or a for-cause biopsy in the Third Post-Transplant Year
Degree of Correlation of Acute Rejection Transcriptional Changes Within the Infiltrating Inflammatory Cells at Year 3 | 3 Years
  Degree Correlation of Transcriptional Changes Within the Infiltrating Inflammatory Cells Assessed by scRNA Sequencing in the Third Post-Transplant Year
Degree of Correlation of Transcriptional Changes Within the Renal Parenchymal Cells at Year 3 | 3 Years
  Degree of Correlation of Acute Rejection Transcriptional Changes Within the Renal Parenchymal Cells Assessed by scRNA Sequencing in the Third Post-Transplant Year
Degree of Correlation of Acute Rejection Transcriptional Changes Within the Infiltrating Inflammatory Cells at year 3 | 3 Years
  Degree of Correlation of Transcriptional Changes Within the Infiltrating Inflammatory Cells of Allograft Biopsy as Assessed by Digital Spatial Transcriptomic Analysis in the Third Post-Transplant Year
Degree of Correlation of Acute Rejection Transcriptional Changes Within the Renal Parenchymal Cells | 3 Years
  Degree of Correlation of Transcriptional Changes Within the Renal Parenchymal Cells with Persistence or Resolution of Allograft Inflammation as Assessed by Digital Spatial Transcriptomic Analysis in the Third Post-Transplant Year

CONTACTS AND LOCATIONS:
Overall Officials: Aravind Cherukuri, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Subject research data/samples may be shared with investigators conducting other research; this information will be shared without identifiable information. Subjects will not be identified in any publication or in the sharing of data about this study.
  These samples and data will be under the control of the listed investigators. Researchers must present a scientifically valid written request to the PI of this study, who will then either approve or deny the request.